CLINICAL TRIAL: NCT04298398
Title: Impact of Mindfulness-Based Cognitive Therapy and Emotion Focused Therapy Group for Cancer Recovery Interventions on Extracellular Vesicles and Psychological Distress in People Who Had Breast, Colorectal or Prostate Cancer: A Preliminary Parallel Randomized Controlled Trial
Brief Title: Impact of Group Psychological Interventions on Extracellular Vesicles in People Who Had Cancer
Acronym: MindGAP-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Portugues de Oncologia, Francisco Gentil, Porto (Other)
Collaborators: Polytechnic Institute of Porto (Other); VTT Technical Research Centre, Finland (Other); University of Oulu (Other); Linnaeus University (Other); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IPO/PI134
Record Dates: First submitted 2020-02-13; First posted 2020-03-06 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Cancer
Keywords: Breast cancer; Prostate cancer; Colorectal cancer; Psychological stress; Anxiety; Depression; Emotion Focused Therapy; Distress; Extracellular vesicles; Exosomes; Biomarkers; Inflammatory response genes; Group interventions; Mindfulness; Mindfulness Based Cognitive Therapy
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Stress, Psychological; Anxiety Disorders; Depression | interventions — Mindfulness-Based Cognitive Therapy; Therapeutics

STUDY DESIGN:
Masking Description: only the investigator responsible for the eligibility assessment would be blind (in the recruitment, in order to assess eligibility to enter the study), before the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness (MBCT) (Experimental): Group therapy based on Mindfulness Based-Cognitive Therapy (MBCT).
  Interventions: Behavioral: Mindfulness Based-Cognitive Therapy (MBCT)
- Emotion Focused Therapy (EFT-CR) (Experimental): Group therapy based on Emotion Focused Therapy for Cancer Recovery (EFT-CR).
  Interventions: Behavioral: Emotion Focused Therapy Group for Cancer Recovery (EFT-CR)
- Control Group (Other): Treatment as Usual is the condition in which participants will follow the usual institutional intervention protocol for medical follow-up and identification, referral and intervention for people identified with significant distress difficulties.
  Interventions: Other: Treatment as usual (no intervention)

INTERVENTIONS:
Behavioral: Mindfulness Based-Cognitive Therapy (MBCT) — MBCT is a program developed by Zindel Segal, Mark Williams and John Teasdale. During MBCT patients learn to decenter their negative thoughts and feelings, allowing the mind to move from an automatic thought pattern to conscious emotional processing. Mindfulness practices included in this program are breath awareness, body scan, sitting and walking meditation, and mindful yoga. The intervention will have the following structure: 8 weekly face-to-face meetings of 2 hours in a group format, daily home-based practice of learned skills, 4 hours of retreat/intensive group work after the fifth week, 6 months of home practice, 4 monthly consolidation face-to-face sessions.
  Arms: Mindfulness (MBCT)
Behavioral: Emotion Focused Therapy Group for Cancer Recovery (EFT-CR) — EFT-CR is an evidence-based approach to psychotherapy, which combines aspects of person-centered, gestalt and existential therapies with contemporary emotion theory and dialectical constructivism (Elliott et al, 2004, Rice & Greenberg, 1984). On EFT-CR, therapist follows the client experience and guides the process, proposing therapeutic tasks when specific client behaviors occur. EFT-CR uses a set of emotion change principles which guide a process of emotional deepening process, from undifferentiated distress to secondary reactive emotions to primary maladaptive emotions to core pain and thence to primary adaptive emotions and emotional transformation (Elliott & Greenberg 2016). The intervention will have the following structure: 8 weekly face-to-face meetings of 2 hours in a group format, daily home-based practice of learned skills, 4 hours of retreat/intensive group work after the fifth week, 6 months of home practice, 4 monthly consolidation face-to-face sessions.
  Arms: Emotion Focused Therapy (EFT-CR)
Other: Treatment as usual (no intervention) — Treatment as Usual is the condition in which participants will follow the usual institutional intervention protocol for medical follow-up and identification, referral and intervention for people identified with significant distress difficulties.
  Arms: Control Group

SUMMARY:
Background: There is some evidence demonstrating the effect of psychological interventions in improvements in health biological parameters. To best of our knowledge, no study had addressed the impact of any psychological intervention on extracellular vesicles. In addition, Mindfulness-Based Cognitive Therapy (MBCT) and Emotion Focused Therapy for Cancer Recovery (EFT-CR) in the group have never been explored regarding extracellular vesicles and the effectiveness of these was not compared yet.

Objectives:

1. To explore and compare the effect of MBCT and EFT-CR on biological parameters and psychological variables in distressed people who have had breast, prostate and colorectal cancer;
2. In addition, we will explore the acceptability through recruitment and retention rates of MBCT and EFT-CR in group and evaluate whether these interventions are appropriate for a larger clinical trial.

Methods: The design of this study is a parallel randomized controlled trial. Participants will be randomized into MBCT, EFT-CR or usual care. Outcome measures will be assessed before, at the end of the intervention (8 weeks) and follow-ups (24 and 52 weeks from the baseline moment).

Hypotheses: The researchers expected that both interventions will have an effect on extracellular vesicles and other study biomarkers as well as improvements in psychological outcomes, compared to treatment as usual (TAU) group. Regarding the comparative effectiveness, we did not have evidence to hypothesize which one of the interventions will be superior in both biological (extracellular vesicles) and psychological outcomes.

Contribution for practice: The results of this preliminary study would permit to know if there are benefits of these psychological interventions on changes in extracellular vesicles and on psychological outcomes related to health. In addition, this study will permit to determine the acceptability of conducting a larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 18 to 65
* Diagnosed with breast, prostate, or colorectal cancer
* Have been diagnosed with cancer stage I-III
* Have finished cancer treatments from 3 months to 2 years (it will be included ongoing hormonal therapies)
* Experiencing significant distress (5 or more) on the Distress Thermometer at baseline
* Available to attend the intervention for the trial duration
* Sufficient functional ability to participate in intervention groups (ECOG)
* Ability to speak and write Portuguese and literacy to autonomous completion of questionnaires

Exclusion Criteria:

* Patients in treatments such as ongoing chemotherapy or radiotherapy, or trastuzumab therapy
* Patients with ostomy
* A diagnosis of a concurrent disorder of psychosis, substance abuse, bipolar disorder, or active suicidality
* Current use of antipsychotics
* Current use of anti-inflammatory medication (corticotherapy)
* Currently engaging in a mindfulness meditation practice or yoga, or having done so within the previous year
* Being under any actual psychosocial or psychological treatment
* Participation in a MBCT program in the last five years
* Pregnancy or breast feeding
* A diagnosis of a concurrent autoimmune disorder

Study Population Description: Participants will be recruited in the Portuguese Oncology Institute of Porto (Porto, Portugal), which is a reference public hospital in the north of the country offering cancer treatments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change on Extracellular vesicles number by ultracentrifugation with sucrose cushion | T0-before intervention; T1-8 weeks after T0; T2-24 weeks after T0; T3-52 weeks after T0
  The collected extracellular vesicles will be quantified by Nanoparticle tracking analysis (Nanosight Ltd.), and data will be measured in particles per milliliter (mL). NTA measures Brownian movements on a particle-by-particle basis tracking movements by image analysis. Additionally, miR21-5p - a brain related microRNA - will be measured to ascertain for the extracellular vesicle's origin. The latter will be achieved by isothermal DNA amplification method, and data will be measured by luminescence (in RLU - relative light unit).
Change on anxiety, depression and stress (Depression Anxiety Stress Scales, DASS21) | T0-before intervention; T1-8 weeks after T0; T2-24 weeks after T0; T3-52 weeks after T0
  This self-report instrument assess the depressive, anxiety and stress symptoms in a 4-points likert scale, from 0 to 3, with higher values representing higher depression, anxiety and stress symptoms

SECONDARY OUTCOMES:
Change on Cancer antigen (CA 15-3) | T0-before intervention;T2-24 weeks after T0; T3-52 weeks after T0
  This indicator assess CA 15-3 (units/mL) using an immunoassay analyzer
Change on Prostate-specific antigen (PSA) | T0-before intervention;T2-24 weeks after T0; T3-52 weeks after T0
  This indicator assess PSA (ng/mL) using an immunoassay analyzer
Change on Carcinoembryonic Antigen assays (CEA) | T0-before intervention;T2-24 weeks after T0; T3-52 weeks after T0
  This indicator assess CEA (ng/mL) using an immunoassay analyzer
Change on Adrenocorticotropic Hormone (ACTH) | T0-before intervention;T2-24 weeks after T0; T3-52 weeks after T0
  This indicator assess ACTH (pg/mL) using an immunoassay analyzer
Transcript inflammatory response genes (IL-1, IL-6, IL-8, IL-10, IFNγ and TNF) | T0-before intervention; T2-24 weeks after T0; T3-52 weeks after T0
  These indicators assess inflammatory response genes in plasma by Quantitative RT-PCR assays of the same individuals using TaqMan™ Gene Expression Assays
Change on Analytic biomarkers (Erythrocytes number) | T0-before intervention; T2-24 weeks after T0; T3-52 weeks after T0
  This indicator assess erythrocytes number (million/mm3) from blood samples(Sysmex XN)
Change on Analytic biomarkers (PCR number) | T0-before intervention; T2-24 weeks after T0; T3-52 weeks after T0
  This indicator assess PCR (mg/L) from blood samples
Change on Analytic biomarkers (telomerase activity) | T0-before intervention; T2-24 weeks after T0; T3-52 weeks after T0
  This indicator assess telomerase activity (units) from blood samples
Change on Analytic biomarkers (hemoglobin glycosylated (HPLC)) | T0-before intervention; T2-24 weeks after T0; T3-52 weeks after T0
  This indicator assess HPLC (mmol/mol) from blood samples
Change on Global distress (Clinical Outcome Routine Evaluation - Outcome Measure, CORE-OM) | T0-before intervention; T1-8 weeks after T0; T2-24 weeks after T0; T3-52 weeks after T0
  This self-report measure assesses global distress in four domains: subjective well-being, symptoms, social/life functioning, risk to self and others, rated in 5-points likert scale from never to always. Higher scores meaning higher psychological suffering
Change on quality of life (Functional Assessment of Cancer Therapy, FACT) | T0-before intervention; T2-24 weeks after T0; T3-52 weeks after T0
  These self-report instrument assess perceived quality of life related to the cancer, in a 5-points likert scale, from 0 to 4, with higher value indicated higher quality of life
Change on quality of life (Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale, FACIT-SP) | T0-before intervention; T2-24 weeks after T0; T3-52 weeks after T0
  These self-report instruments assess perceived spiritually related to the cancer in a 5-points likert scale, from 0 to 4, with higher value indicated higher well-being
Change on fear of cancer recurrence (Fear of Cancer Recurrence, FCR-7) | T0-before intervention; T1-8 weeks after T0; T2-24 weeks after T0; T3-52 weeks after T0
  This self-report instrument assess the fear of cancer recurrence, rated in a 5-points likert scale, with higher values indicated higher fear of recurrence
Change on satisfaction perceived social support (ESSS) | T0-before intervention; T1-8 weeks after T0; T2-24 weeks after T0; T3-52 weeks after T0
  This self-report instrument assess the perceived level of social support, rated in a 5-points likert scale, with higher values meaning higher social support
Change on emotional regulation processes (Emotion Regulation Questionnaire, ERQ, emotion suppression subscale) | T0-before intervention; T1-8 weeks after T0; T2-24 weeks after T0; T3-52 weeks after T0
  This self-report measure assess the emotion regulation processes rated in a 7-points likert scale, with higher values representing higher emotional suppression
Change on impact of events (Impact of Event Scale - Revised, IES-R) | T0-before intervention; T1-8 weeks after T0; T2-24 weeks after T0; T3-52 weeks after T0
  This self-report measure assess the impact of significant events, rated in a 5-points likert scale, with higher scores meaning higher negative impact of the event
Change on Mindfulness Attention and Awareness (Mindfulness Attention and Awareness Scale, MAAS) | T0-before intervention; T1-8 weeks after T0; T2-24 weeks after T0; T3-52 weeks after T0
  This self-report measure assess the mindfulness and awareness skills, rated in a 6-points likert scale with higher scores indicating higher attention and awareness
Change on self-compassion skills (Self-Compassion Scale - Short Form, SHORT FORM) | T0-before intervention; T1-8 weeks after T0; T2-24 weeks after T0; T3-52 weeks after T0
  This self-report measure assess the self-compassion skills, rated in 5-points likert scale, with higher scores indicating higher self-compassion
Change Interview (Elliot, 1999) | T2-24 weeks after T0
  This interview assesses the psycho-therapeutic changes perceived by participants after psychological intervention. The interview questions explore the changes that a person has noticed since therapy began, what the person attributes these changes to, and helpful and unhelpful aspects of therapy, in a qualitative way. In addition, the participants identified therapeutic changes as result of the therapy and are asked to rate these changes in three scales: expected change (1: change totally expected; 5: totally unexpected); change without therapy (1: the change would not have happened; 5: change would happen for sure); and the value of the change (1: nothing important; 5: extremely important).
Change on smoking dependency (Fagestrom Test) | T0-before intervention; T2-24 weeks after T0; T3-52 weeks after T0
  This instrument assesses nicotine dependency with 6 items (rated from 0 to 2 or 3). The total score range is 1-10, with higher values meaning higher nicotine dependency
Change on physical activity (IPAQ,The International Physical Activity Questionnaire) | T0-before intervention; T2-24 weeks after T0; T3-52 weeks after T0
  This instrument assesses physical activity in 7 items, with higher scores meaning higher level of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Rui Henrique, PhD, Study Chair — IPO-Porto; Carmen Jerónimo, PhD, Study Director — IPO-Porto; Eunice Silva, PhD, Study Director — IPO-Porto; Goreti Sales, PhD, Study Director — ISEP-Biomark (Polytecnic Institute of Porto)